CLINICAL TRIAL: NCT05363280
Title: A Phase 2 Evaluation of the Safety and Efficacy of AL8326 in ≥2nd Line Small Cell Lung Cancer (SCLC) Treatment
Brief Title: Phase 2 Safety and Efficacy Evaluation of AL8326 in ≥2nd Line SCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Advenchen Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Organization: Advenchen Laboratories, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL8326-US-001
Record Dates: First submitted 2022-04-22; First posted 2022-05-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Small Cell Lung Cancer
Keywords: Recurrent small cell lung caner; Advanced small cell lung cancer; Metastatic Small lung cancer; ≥2nd Line treatment
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The phase 2 study aims to find optimal biological dose (OBD) for Phase 2 expansion cohort clinical study. Patients will be randomized to a 3 different dosing daily AL8326 groups ( low. middle. high) in 1:1:1 ratio in OBD finding cohorts.
  A phase 2 expansion cohort will be continued if a positive clinical result would have been observed after OBD determination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- OBD finding cohort at low dose (Experimental): Subject in low dose group will receive AL8326 orally in each cycle until intolerable toxicity or disease progression or withdrawal . 6-12 subjects are in this group. Efficacy, safety and PK will be evaluated and compared within 3 different dosing group to define the final OBD.
  Interventions: Drug: AL8326 low dose group
- OBD finding cohort at middle dose (Experimental): Subject in middle dose group will receive AL8326 orally in each cycle until intolerable toxicity or disease progression or withdrawal . 6-12 subjects are in this group. Efficacy, safety and PK will be evaluated and compared within 3 different dosing group to define the final OBD.
  Interventions: Drug: AL8326 middle dose group
- OBD finding cohort at high dose (Experimental): Subject in high dose group will receive AL8326 orally in each cycle until intolerable toxicity or disease progression or withdrawal . 6-12 subjects are in this group. Efficacy, safety and PK will be evaluated and compared within 3 different dosing group to define the final OBD.
  Interventions: Drug: AL8326 high dose group

INTERVENTIONS:
Drug: AL8326 low dose group — Taken AL3826 at low dose orally
  Arms: OBD finding cohort at low dose
Drug: AL8326 middle dose group — Taken AL3826 at middle dose orally
  Arms: OBD finding cohort at middle dose
Drug: AL8326 high dose group — Taken AL3826 at high dose orally
  Arms: OBD finding cohort at high dose

SUMMARY:
This trial is a Phase II trial designed to evaluate the safety and efficacy of using oral AL8326 , a multi-targeted receptor Tyrosine Kinase Inhibitor( TKI) , to recurrent, advanced, or metastatic small cell lung cancer (SCLC) patients who need ≥2nd line treatment .

DETAILED DESCRIPTION:
This study is designed for two steps: Phase 2 Optimal Biological Dose (OBD) finding and Phase 2 expansion cohort study after OBD determination.

The Phase 2 study aims to find optimal biological dose (OBD) initially. Patients will be randomized to 3 different dosing groups in OBD finding cohorts. Each cohort will enroll 6-12 SCLC patients who need ≥2nd line treatment without or with brain metastasis which is controlled with no active hemorrhage. This OBD finding cohort will also evaluate the pharmacokinetic profile of AL8326.

A phase 2 expansion cohort will be continued if a positive clinical result would have been observed after OBD determination for 40-60 patients. Upon FDA's approval the Phase 2 expansion cohort clinical study will be further expanded to evaluate the safety and efficacy of AL8326 in patients individually with SCLC who need = or >2nd line treatment without or with brain metastasis which is controlled with no active hemorrhage.

ELIGIBILITY:
Major Inclusion Criteria:

1. Male or female, 18 years of age or older
2. ECOG performance status of 0 or 1
3. Histologically or cytologically confirmed SCLC
4. Have at least 1 lesion that meets the criteria for being measurable, as defined by RECIST 1.1
5. Have a life expectancy of at least 3 months

Major Exclusion Criteria:

1. Serious, non-healing wound, ulcer or bone fracture
2. Major surgical procedure within 28 days or minor surgical procedure performed within 7 days prior to treatment
3. Active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
4. Clinically significant cardiovascular disease including uncontrolled hypertension; myocardial infarction or unstable angina within 6 months prior to enrollment; New York Heart Association (NYHA) Grade II or greater congestive heart failure serious cardiac arrhythmia requiring medication; and Grade II or greater peripheral vascular disease
5. Hemoptysis within 3 months prior to enrollment
6. Concomitant treatment with strong inhibitors or inducers of CYP3A4, CYP2C9 and CYP2C19 within 14 days prior to enrollment and during the study unless there is an emergent or life-threatening medical condition that required it.

More information available upon request

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Optimal biological dose ( OBD ) | 12 months
  Determine the Optimal biological dose ( OBD ) via evaluation of dose limiting toxicity (DLT) events to decide the dosing using in expanded cohort
Objective Response Rates (ORR) | 12 month
  Evaluate the efficacy among 3 different dosing groups

SECONDARY OUTCOMES:
Duration of response ( DOR) | 12 months
  Measure the length of time that a tumor continues to respond to treatment without the cancer growing or spreading
Number of participants with AEs, SAEs, abnormal physical examination findings, abnormal laboratory test results, abnormal vital signs and abnormal electrocardiography (ECG) findings | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Saiama Waqar, MD, Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Siteman Cancer Center, Washington University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramón Y Cajal, Madrid